CLINICAL TRIAL: NCT07269795
Title: Advanced Strategy of Food Supplements for the Optimization of Satiety and Lipid Metabolism in Maturity
Brief Title: Advanced Strategy of Food Supplements for the Optimization of Satiety and Lipid Metabolism in Maturity (SACIANS)
Acronym: SACIANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, Prof. Dr. Alejandro Martínez-Rodríguez, Catedrático Ciencias de la Salud, University of Alicante
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UA-2025-04-15
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Dyslipidemia; Lipid Metabolism; Satiety Response; Overweight and/or Obesity
Keywords: Food supplements; Satiety; Lipid metabolism; Overweight; Middle-aged adults; Metabolic health; Nutraceuticals; Mediterranean diet; Body composition
MeSH Terms: conditions — Dyslipidemias; Overweight

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: a control group (no supplementation) and an intervention group (receiving the supplement combination). Both groups will follow their habitual diet and lifestyle during the 12-week intervention.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to group allocation during data analysis to minimize bias. Given the nature of the intervention (supplementation vs. no supplementation), participant blinding is not applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group - Food Supplement Combination (Experimental): Participants in this group will receive a daily combination of commercially available food supplements for 12 weeks.
  The selection of supplements will be based on safety criteria, nutritional labeling, and prior evidence of beneficial effects on satiety and lipid metabolism.
  The supplements are registered as food supplements available in pharmacies and herbal stores.
  Participants will maintain their habitual diet and lifestyle throughout the study period.
  Interventions: Dietary Supplement: Food Supplement Combination (SACIANS Formula)
- Control Group - No Supplementation (No Intervention): Participants in this group will not receive any supplementation during the 12-week study period.
  They will maintain their usual diet and lifestyle, serving as the control group for comparison with the experimental supplementation group.

INTERVENTIONS:
Dietary Supplement: Food Supplement Combination (SACIANS Formula) — Participants in the experimental group will receive a combination of commercially available food supplements daily for 12 weeks.
  The specific supplements will be selected based on safety, labeling accuracy, and prior evidence of beneficial effects on satiety and lipid metabolism.
  All supplements are registered as food supplements and are commercially available in pharmacies and herbal stores.
  The combination aims to enhance satiety, improve lipid metabolism, and promote metabolic health in overweight adults.
  Participants will be instructed to maintain their usual diet and lifestyle habits throughout the intervention period.
  Arms: Experimental Group - Food Supplement Combination

SUMMARY:
The SACIANS study (Advanced Strategy of Food Supplements for the Optimization of Satiety and Lipid Metabolism in Middle-Aged Adults) aims to evaluate the combined effect of commercially available food supplements on satiety and lipid metabolism in adults over 45 years of age who are overweight.

This 12-week randomized controlled clinical trial will include 80 participants divided into two parallel groups: a control group without supplementation and an experimental group receiving a specific combination of food supplements with proven nutritional safety and previous evidence of functional effects on metabolism.

Primary outcomes include changes in biochemical parameters related to lipid metabolism (cholesterol profile, triglycerides, and glucose), as well as markers of oxidative stress and inflammation. Secondary outcomes include variations in body composition, perceived satiety, emotional well-being, sleep quality, and lifestyle habits such as diet adherence and physical activity.

The study will be conducted at the University of Alicante and the EIEH Clinic (Elche Institute of Exercise and Health), following the principles of the Declaration of Helsinki. The goal is to provide scientific evidence on the synergistic potential of existing food supplement combinations to promote metabolic balance and healthy aging.

DETAILED DESCRIPTION:
Overweight and metabolic alterations in adults over 45 years old represent a growing public health concern, frequently associated with conditions such as type 2 diabetes, dyslipidemia, and cardiovascular disease. Although numerous food supplements are currently available on the market with reported effects on satiety or lipid oxidation, most lack personalization and evidence regarding their combined effects.

The SACIANS project (Advanced Strategy of Food Supplements for the Optimization of Satiety and Lipid Metabolism in Middle-Aged Adults) is a 12-week, randomized, controlled, parallel-group clinical trial designed to evaluate the efficacy of different combinations of commercially available food supplements on metabolic and emotional parameters in adults with overweight or mild obesity.

Participants (n = 80; 40 per group) will be randomly assigned to one of two arms:

Control group: No supplementation.

Experimental group: Daily intake of a combination of registered food supplements selected based on their nutritional profile, labeling, safety, and prior evidence of functional efficacy.

Assessments will include biochemical parameters (glucose, lipid profile, oxidative and inflammatory biomarkers), body composition (via bioimpedance and 3D scanning), blood pressure, and psychological well-being (stress, anxiety, and sleep quality). Lifestyle factors such as Mediterranean diet adherence and physical activity (recorded with Fitbit) will also be monitored.

The trial will follow the ethical standards of the Declaration of Helsinki and has been approved by the Ethics Committee of the University of Alicante (approval date: May 29, 2025). Statistical analyses will be performed using SPSS v24.0, applying repeated-measures ANOVA and appropriate post hoc corrections.

This study aims to identify potential synergistic effects among existing food supplement formulations, contributing to the rational and evidence-based use of these products for improving satiety, lipid metabolism, and metabolic health in adults.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years
* Body Mass Index (BMI) between 25.0 and 34.9 kg/m²
* Signed informed consent form

Exclusion Criteria:

* Pregnancy or breastfeeding
* Participation in similar studies within the previous 3 months
* Current use of supplements or medications that may affect metabolism
* Joint injury or physical limitation that restricts participation
* Clinical conditions that could prevent adherence to the study protocol

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Change in total cholesterol | Baseline and after 12 weeks of intervention
  Variation in plasma total cholesterol concentration after 12 weeks of supplementation.
Change in LDL-cholesterol | Baseline and after 12 weeks of intervention
  Variation in low-density lipoprotein (LDL) cholesterol levels to evaluate lipid metabolism response.
Change in perceived satiety levels | Baseline and after 12 weeks of intervention
  Evaluation of subjective satiety using a validated visual analog scale (VAS) for appetite and fullness.
Change in HDL-cholesterol | Baseline and after 12 weeks of intervention
  Variation in high-density lipoprotein (HDL) cholesterol levels as an indicator of cardiovascular health.
Change in triglycerides | Baseline and after 12 weeks of intervention
  Variation in plasma triglyceride concentration
Change in fasting glucose | Baseline and after 12 weeks of intervention
  Difference in fasting blood glucose concentration after the intervention period.

SECONDARY OUTCOMES:
Change in body weight | Baseline and after 12 weeks of intervention
  Change in total body weight measured using a calibrated scale.
Change in body fat percentage | Baseline and after 12 weeks of intervention
  Variation in body fat percentage measured by 3D body scan (SCANECA).
Change in lean mass | Baseline and after 12 weeks of intervention
  Difference in lean body mass determined by bioimpedance and 3D body scan (SCANECA).
Change in C-reactive protein (CRP) | Baseline and after 12 weeks of intervention
  Variation in serum CRP concentration as a marker of systemic inflammation
Change in malondialdehyde (MDA) | Baseline and week 12
  Difference in plasma MDA concentration as an oxidative stress biomarker
Change in total antioxidant capacity (TAC) | Baseline and week 12
  Variation in total antioxidant capacity of plasma
Change in perceived stress (PSS questionnaire) | Baseline and week 12
  Range: 0-40. Interpretation: Higher scores indicate greater perceived stress. Description: The PSS-10 is a 10-item self-reported questionnaire that measures the degree to which situations in one's life are appraised as stressful during the past month. Items are rated on a 5-point Likert scale (0 = never to 4 = very often). Scores are summed to obtain a total perceived stress score, where higher values reflect greater stress perception.
Change in sleep quality (PSQI) | Baseline and week 12
  Range: 0-21. Interpretation: Higher scores indicate worse sleep quality. Description: The PSQI is a self-reported questionnaire that assesses sleep quality and disturbances over a 1-month period. It consists of 19 items grouped into seven components (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction), each scored 0-3. The sum of the components yields a global score (0-21).
Change in Mediterranean diet adherence (PREDIMED score) | Baseline and week 12
  Range: 0-14. Interpretation: Higher scores indicate better adherence to the Mediterranean diet. Description: The PREDIMED questionnaire evaluates adherence to the Mediterranean dietary pattern through 14 items covering key aspects such as olive oil intake, fruit and vegetable consumption, fish intake, and limited consumption of red meat and sweets. Each affirmative answer scores 1 point.
Change in physical activity level (IPAQ questionnaire) | Baseline and week 12
  Range: 0 to unlimited MET-min/week (commonly categorized into 3 levels: low, moderate, high). Interpretation: Higher scores indicate higher levels of physical activity. Description: The IPAQ-SF measures physical activity over the last 7 days through 7 items that estimate the time spent walking, and performing moderate and vigorous activities. Results are expressed in MET-minutes per week or categorized according to intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- European Institute Of Exercise and Health, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No